CLINICAL TRIAL: NCT00436371
Title: The Use of Amisulpride in Schizophrenic Acute Phase Patients.
Brief Title: Amisulpride in Schizophrenic Acute Phase Patients
Acronym: ASAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9517
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride

ARMS (1):
- 1 (Experimental): Amisulpride 400-800mg per day on a twice-a-day regimen
  Interventions: Drug: Amisulpride

INTERVENTIONS:
Drug: Amisulpride — Oral tablets

SUMMARY:
To collect the safety and response of using Amisulpride in acute schizophrenic patients

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed as Diagnostic and Statistical Manual of Mental Disorder, 4th edition, as paranoid, disorganized or undifferentiated type of schizophrenia in acute episode

Exclusion Criteria:

* Patients previously treated with amisulpride
* Patients have comorbidity which may interfere with the treatment or follow-up
* Patients currently taking depot antipsychotics (at least 30 days washout period is needed)
* Patients currently/ or recently (< 3 months) withdrawn from drug or alcohol abuse
* Pregnant or lactation

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-05; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | all across the study

SECONDARY OUTCOMES:
Clinical Global Impressions | All accross the study
Patient compliance | all across the study
Percentage of patient completing treatment | all across the study
Changes in body weight | At baseline and day 84

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Tang, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Hong Kong, Hong Kong